CLINICAL TRIAL: NCT05454514
Title: Automated Medication Platform With Video Observation and Facial Recognition to Improve Adherence to Antiretroviral Therapy in Patients With HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Gellman (Industry)
Responsible Party: Sponsor-Investigator, Charles Gellman, PI, HiDO Technologies
Organization: HiDO Technologies (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R43MH125483-01A1 (NIH)
Record Dates: First submitted 2022-07-02; First posted 2022-07-12 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: HiDO is an automated Artificial Intelligence driven direct observation medication adherence platform. The platform is a 510K exempt Class I medical device that integrates medication dispensing, dose administration time, pill count and front facing video cameras to validate the right medications, at right time to the right patient. The device dispenses up to 7 different types of medications simultaneously. The camera logs every dose using facial recognition and provides real time consumption logs. Investigators have access to video observation logs, patient dose time, adherence trends, and study level adherence measures.
Masking Description: This is a randomized, unblinded, Phase 1 study of the HiDO automated medication adherence platform in patients ages 18 to 65 with HIV/AIDS who are currently taking ART. For this single-site device study, clinical collaborators will recruit 24 subjects into a single study group. After a screening period of up to 14 days, subjects will receive the 90-day intervention that consists of using of an automated medication adherence platform. Medication adherence will be assessed through observed therapy using front-facing cameras on the device. Corroborating data will be drawn from viral load data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Automated Medication Platform with Video Observation (Other): There is no drug intervention. The device elicits increases adherence of medications.
  Interventions: Device: HiDO medication adherence platform; Device: Automated Medication Platform with Video Observation; Other: Time on Task

INTERVENTIONS:
Device: HiDO medication adherence platform — The HiDO medication adherence platform will be shipped directly to the home of record of each participant. The Primary Endpoint is medication adherence as assessed by remote observation through the HiDO device at 90 days.
Device: Automated Medication Platform with Video Observation — There is no drug intervention. The device elicits increases adherence of medications.
Other: Time on Task — Other Endpoints include Time on Task for initial registration, "first click" testing, facial recognition setup, medication administration, number and type of critical and non-critical errors and error-free rate, System Usability Scale (SUS), and Net Promoter Score.

SUMMARY:
This is a 90-day medication adherence study testing the HiDO is an automated AI-driven direct observation medication adherence platform, which is a 510K-exempt, Class I medical device with 24 people with HIV/AIDS, ages 18 to 55, who are currently taking ART and reporting less than 100% adherence. The aims of the study are to see whether the device can achieve >95% ART adherence among all participants averaged over 90 days and to perform usability testing using the System Usability Scale and Net Promoter scores.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) is directly responsible for reducing the death rate from HIV/AIDS. AIDS-related deaths declined by 38% from 2000 to 2017-saving more than 11 million lives worldwide. Mediation adherence is critically important to this statistic and to clinical trials. Investigators insist on (or assume) adherence rates of ≥95%. However, when bodily fluid measurements are used to assess adherence, the values are substantially lower: 54% to 68%. Viral suppression generally requires most ART be taken with at least 95% adherence. Poor adherence to ART during a clinical trial can underestimate efficacy, increase subject discontinuation rates, and extend recruitment periods and the total duration of clinical trials. This is expensive for clinical trial sponsors and slows or halts the development of antiretrovirals. Direct observation is the gold standard for medication adherence but is prohibitively expensive and impractical. HiDO is an automated AI-driven direct observation medication adherence platform. The platform is a 510K-exempt, Class I medical device with a provisional patent that integrates medication dispensing, pill count and a front-facing video cameras to confirm the right medications are given at right time to the right patient. Investigators have access to video observation logs, patient dose time, adherence trends, and study-level adherence through the platform's dashboard. Data is stored securely in the cloud and accessible real-time. The device dispenses up to 7 different types of medications simultaneously, 40 doses each. During the 90-day study, participants will receive smart phone reminders; pills will be dispensed through the unit and adherence monitored and verified through video observation and facial recognition. Our benchmark for success is that all participants who complete the study will achieve ≥95% adherence to ART averaged across 90 days (Milestone 1). Adherence will be quantified as the (no. of doses provided - no. of doses taken) / the no. of doses provided X 100. The investigators will further confirm adherence by reviewing patient charts for viral load and CD4 T-cell count. In the same study population described above, the investigators will conduct full usability testing at 2 weeks of use. The investigators will measure Time on Task for initial registration, "first click" testing, facial recognition setup, and medication administration, and assess the number and type of critical and non-critical errors and error-free rate. Results of usability testing will be equal to or better than published benchmark rates for similar platforms (Milestone 2). Subjects will complete the 10-item System Usability Scale (SUS) and achieve an average SUS score >68 (Milestone 3). More than 80% of subjects will have Likely or Strongly Likely Net Promoter Score (Milestone 4). If successful, the investigators will have demonstrated that our automated medication adherence platform is highly usable and user-friendly, enables strict adherence to ART trials, and is ready for testing in Phase II.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Prescription for at least one existing ART
* Has expressed difficulty with medication adherence (question screen)
* Access to a personal smart phone and a Wi-Fi connection
* Ability to read and write English

Exclusion Criteria:

* Illicit drug use within the past 6 months (excl. marijuana)
* Diagnosis of dementia
* Clinical study participation within the previous 3 months
* Changes to ART regimen within the previous 2 months
* Anticipated change to ART therapy within the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HiDO Technologies Inc., El Dorado Hills, California, United States

IPD SHARING:
Plan to Share IPD: No
Results will not be published.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study successfully recruited 7 patients with HIV/AIDS who met the inclusion criteria, which include age between 18-55, existing prescription for at least one ART, expressed difficulty with medication adherence, access to a personal smartphone and Wi-Fi connection, and the ability to read and write English.To ensure unbiased and rigor results, the inclusion criteria was confirmed by the study team.
Groups:
- Automated Medication Platform With Video Observation: There is no drug intervention. HiDO medication adherence platform: The device elicits increases adherence of medications. The Primary Endpoint is medication adherence as assessed by remote observation through the HiDO device at 90 days. Time on Task: Other Endpoints include Time on Task for initial registration, "first click" testing, facial recognition setup, medication administration, number and type of critical and non-critical errors and error-free rate, System Usability Scale (SUS), and Net Promoter Score.
Period: Overall Study
Arm/Group | Automated Medication Platform With Video Observation
Started | 7
Completed | 3
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: The study collected self-reported adherence data during screening, recognizing that while patients tend to overestimate adherence, those admitting to taking less than 100% of ART doses in the past 30 days were accurately reporting suboptimal adherence. This self-report served as a baseline for comparison to later adherence measurements.
Groups:
- Automated Medication Platform With Video Observation: There is no drug intervention. HiDO medication adherence platform: The device elicits increases adherence of medications.
Arm/Group | Automated Medication Platform With Video Observation
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Medication Adherence
Description: The primary endpoint was to determine the number of participants who achieved 80-95% adherence to ART medications averaged across 90 days (Milestone 1). The benchmark for success was set at all participants completing the study achieving adherence within this range. Adherence rates were calculated as the number of doses provided minus the number of doses missed, divided by the total number of doses provided, multiplied by 100.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Automated Medication Platform With Video Observation
Number analyzed (Participants) | 3
Participants
  Percentage of adherence ≥95% adherence | 2
  Number/Percentage of participants with 80% to 95% adherence. | 1

ADVERSE EVENTS:
Time Frame: Participants in this study were assessed over a 90-day intervention period.
Description: Adverse events (AEs) were monitored throughout the 90-day study. Serious adverse events (SAEs) were defined per MedDRA 10.0 and reported to the Safety Review Committee within 24 hours. Non-serious AEs were documented and tracked by research coordinators.
Arm/Group | Automated Medication Platform With Video Observation
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT05454514/Prot_SAP_ICF_002.pdf